CLINICAL TRIAL: NCT02654652
Title: Intestinal Function of Patients With Uper Air and Digestive Neoplasia Submitted to Surgical Treatment: Symbiotic Use Impact
Brief Title: Impact of Symbiotic Administration on Intestinal Function of Head and Neck Patients Surgically Treated
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CAAE 24375713.0.0000.5149
Record Dates: First submitted 2016-01-07; First posted 2016-01-13 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-02

CONDITIONS: Head and Neck Cancer; Synbiotics; Nutrition Therapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symbiotic (Experimental): Patients will receive the symbiotic product LactoFos twice a day during seven days after surgical treatment. The intervention consists of giving twice a day a sachet of 6g of symbiotic diluted in 20mL of water via nasoenteric tube for seven days, totaling the administration of 14 sachets per intervention.
  Interventions: Dietary Supplement: Symbiotic
- Maltodextrin (Placebo Comparator): Patients will receive 6g of maltodextrin twice a day during seven days after surgical treatment.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Symbiotic — Intervention will consist of the adminitration of symbiotic product twice a day during seven days after surgical treatment
  Other Names: LactoFos
  Arms: Symbiotic
Dietary Supplement: Maltodextrin — Intervention will consist of the adminitration of placebo product twice a day during seven days after surgical treatment
  Arms: Maltodextrin

SUMMARY:
The purpose of this study is to determine whether the symbiotic use in patients with head and neck cancer impact on intestinal function after surgical treatment.

DETAILED DESCRIPTION:
The study will be conducted offering the patients symbiotic product twice a day for seven days after the surgical treatment. Patients will be monitored for the number of stools, stools consistency, abdominal pain and gas overproduction.

ELIGIBILITY:
Inclusion Criteria:

* head and neck cancer with primary surgical treatment, enteral nutrition by enteral tube.

Exclusion Criteria:

* three months antibiotic use earlier the surgery, recently radiotherapy or quimiotherapy, inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla C Lages, bachelor, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- UFMG Hospital, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Result] Detsky AS, McLaughlin JR, Baker JP, Johnston N, Whittaker S, Mendelson RA, Jeejeebhoy KN. What is subjective global assessment of nutritional status? 1987. Classical article. Nutr Hosp. 2008 Jul-Aug;23(4):400-7. No abstract available. PMID 18702178
- [Derived] Lages PC, Generoso SV, Correia MITD. Postoperative symbiotic in patients with head and neck cancer: a double-blind randomised trial. Br J Nutr. 2018 Jan;119(2):190-195. doi: 10.1017/S0007114517003403. Epub 2017 Dec 26. PMID 29277158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients hospitalized with head and neck cancer from Instituto Alfa de Gastroenterologia, Hospital das Clínicas de Minas Gerais, from October 2014 until April 2016
Pre-assignment Details: Of the 40 patients screened, six were ineligible: esophageal cancer (1), cirrhosis (1) and four were inoperable. Forty were randomized (19 - symbiotic group and 21 - control)
Groups:
- Symbiotic: Patients will receive twice a day the symbiotic product during seven days after surgical treatment
  LactoFos: Patients will receive the product twice a day during seven days after surgical treatment
- Maltodextrin: Patients will receive twice a day the placebo product during seven days after surgical treatment
  Maltodextrin: Patients will receive maltodextrin twice a day during seven days after surgical treatment
Period: Overall Study
Arm/Group | Symbiotic | Maltodextrin
Started | 19 | 21
Completed | 18 | 18
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Symbiotic: Patients received, twice a day, the symbiotic product (LactoFos) for at least 5 days and the maximum of 7 days.
- Maltodextrin: Patients will receive twice a day the placebo product (Maltodextrin) or at least 5 days and the maximum of 7 days.
- Total: Total of all reporting groups
Arm/Group | Symbiotic | Maltodextrin | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 6 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 13 | 16 | 29
Nutritional status [Count of Participants; unit: Participants] — According to Detsky et al, 1987
  Participants
    Nourished | 6 | 8 | 14
    Malnourished | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Serum DAO Enzyme Concentration
Description: The intestinal permeability using serum DAO enzyme concentration (ng/mL) was determined by sandwich enzyme-linked immunosorbent assay (ELISA) kit (SEA656Hu), according to Cloud-Clone Corporation® (Huston, TX) specifications.
Time Frame: 7 days
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Symbiotic | Maltodextrin
Number analyzed (Participants) | 18 | 18
ng/mL | 3 [0 to 7] | 2.5 [0 to 6]

2. Secondary Outcome: Infection Rate
Description: According to Dindo et al, 2004
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Symbiotic | Maltodextrin
Number analyzed (Participants) | 18 | 18
Participants | 11 | 7

ADVERSE EVENTS:
Time Frame: 30 days
Description: All-cause Mortality
Arm/Group | Symbiotic | Maltodextrin
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No